CLINICAL TRIAL: NCT05267223
Title: Experience of Physical and Vocational Rehabilitation Amongst Individuals With Paraplegia
Brief Title: Experience of Rehabilitation Amongst Individuals With Paraplegia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Other Study IDs: MMDU/IEC/2154
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Spinal Cord Injuries
Keywords: qualitative research; paraplegia; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Paraplegia: After screening the participants according to the inclusion/exclusion criteria, informed consent will be obtained from all the selected participants. Their demographic details will be obtained and asked for their comfortable time for the interview. Data will be collected by in-depth face to face, semi- structured interviews. Audio/video recording of the interview will be taken & it will be written in English and will be transcribed verbatim also manual notes will be prepared for their analysis after the interview is conducted
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews — Semi-structured interviews with individuals with paraplegia

SUMMARY:
This study is a qualitative study exploring the facilitators to physical and vocational rehabilitation and also explores the barriers in empowering individuals with paraplegia

DETAILED DESCRIPTION:
Spinal cord injury is one of the most distressing medical conditions being encountered by today's health care system. In India incidence of Spinal cord injury accounts for 20 per million per years population with 20,000 cases added every year. Rehabilitation services are of utmost importance in empowering these individuals. So there is a need for more qualitative studies through which needs in rehabilitation services can be upgraded. The aim of the study is to explore the experience of physical and vocational rehabilitation amongst the individuals with paraplegia in India

ELIGIBILITY:
Inclusion Criteria:

* Traumatic & Non-Traumatic paraplegics Both male & female above 18 yrs of age Time since injury of minimum 6 months Community dwelling paraplegics

Exclusion Criteria:

* Communication problems Psychiatric problems or co morbidities like head injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Traumatic & non-traumatic paraplegics having atleast 6 months of time since injury and are community dwelling so that their obstacles in community integration can be noted
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Semi-structured interview | 30minutes-45 minutes
  Semi-structured interview with audio/video recording

CONTACTS AND LOCATIONS:
Overall Officials: AKANKSHA SAXENA, MPT, Principal Investigator — MAHARISHI MARKANDESHWAR INSTITUTE OF PHYSIOTHERAPY & REHABILITATION
Locations (1):
- Maharishi Markandeshwar institute of Medical Sciences and Research, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No